CLINICAL TRIAL: NCT05164978
Title: DEP Combine With PD-1 Antibody as an Treatment for EBV Associated Hemophagocytic Lymphohistiocytosis (HLH)
Brief Title: DEP Combine With PD-1 Antibody as an Treatment for EBV-HLH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Department of Hematology, Beijing Friendship Hospital, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEP,PD-1, HLH
Record Dates: First submitted 2021-06-24; First posted 2021-12-21 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Hemophagocytic Lymphohistiocytosis
Keywords: Hemophagocytic Lymphohistiocytosis; DEP; PD-1 antibody
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic

STUDY DESIGN:
Intervention Model Description: All patients with EBV- HLH receive DEP combine with PD-1 antibody as an treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DEP combine with PD-1 antibody (Experimental): doxorubicin (doxorubicin hydrochloride liposome injection) 25 mg/m2 day 1; etoposide 100 mg/m2 was administered day1; methylprednisolone 1.5mg/kg days 1 to 3,then 0.25mg/kg day 4 to 14; sintilimab injection 200mg day 4. This regimen was repeated after 2 weeks.
  Interventions: Drug: DEP combine with PD-1 antibody

INTERVENTIONS:
Drug: DEP combine with PD-1 antibody — Doxorubicin hydrochloride liposome injection 25 mg/m2 day 1 Etoposide 100 mg/m2 day1 Methylprednisolone 1.5 mg/kg days 1 to day 3, 0.25mg/kg days 4 to 14 Sintilimab Injection 200mg d4
  Other Names: DEP+PD-1

SUMMARY:
This study aimed to investigate the efficacy and safety of DEP (liposomal doxorubicin, etoposide and methylprednisolone) together with PD-1 antibody as an treatment for EBV associated hemophagocytic lymphohistiocytosis.

DETAILED DESCRIPTION:
PD-1 antibody added to the DEP regimen （with or without asparaginases） in EBV-HLH,

ELIGIBILITY:
Inclusion Criteria:

1. Meet hemophagocytic lymphohistiocytosis (HLH)-04 diagnostic criteria; EBV-DNA in peripheral blood or EBER in tissue were positive, patients were diagnosed with EBV associated HLH (EBV-HLH).
2. . The expected survival time is more than 1 month.
3. Age >18 years old, gender is not limited.
4. Serum creatinine ≤ 1.5 times normal；
5. Serum human immunodeficiency virus(HIV) antigen or antibody negative； Hepatitis C virus (HCV) antibody is negative, or HCV antibody is positive, but HCV RNA is negative；HBV copies less than 1E+03 copies/ml.
6. No thyroid dysfunction. The left ventricular ejection fraction (LVEF) was normal.
7. No uncontrollable infection.
8. Contraception for both male or female.

8. Informed consent obtained.

Exclusion Criteria:

1. Allergic to doxorubicin, etoposide and sintilimab Injection
2. Serious immunoreaction: myocardial damage, hepatitis, pneumonia
3. Central nervous system symptoms
4. Serious mental illness;
5. Central nervous system symptoms
6. Serious mental illness;
7. Accumulated dose of doxorubicin above 300mg/m2 or epirubicin above 450mg/m2；
8. Pancreatitis history. Patients unable to comply during the trial and/or follow-up phase;
9. Participate in other clinical research at the same time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of treatment response | Change from before and 2,4,6 and 8 weeks after initiating DEP combine with PD-1 antibody therapy
  The primary observed endpoint is the objective remission rate (ORR): cases that include complete remission (CR) and partial remission (PR).CR was defined as normalization of all of the quantifiable symptoms and laboratory markers of HLH, including levels of sCD25, ferritin, and triglyceride; hemoglobin; neutrophil counts; platelet counts; and alanine aminotransferase (ALT). PR was defined as at least a 25% improvement in 2 or more quantifiable symptoms and laboratory markers as follows: sCD25 response was>1.5-fold decreased; ferritin and triglyceride decreased at least 25%; for patients with an initial neutrophil count of<0.5 ×109/L, a response was defined as an increase by at least 100% to>0.5× 109/L; for patients with a neutrophil count of 0.5 to 2.0 × 109/L, an increase by at least 100% to >2.0 × 109/L was considered a response; and for patients with ALT >400 U/L, response was defined as an ALT decrease of at least 50%.

SECONDARY OUTCOMES:
EBV-DNA | Change from before and 2,4,6 and 8 weeks after initiating DEP combine with PD-1 antibody therapy
  EBV-DNA copies/ml in peripheral blood
Survival | 3 months after the intervention
  Outcome of patients with EBV-HLH
Adverse events that are related to treatment | 2,4,6 and 8 weeks after initiating DEP combine with PD-1 antibody therapy
  Incidence of events that are related to treatment including myelosuppression, infection, bleeding and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Wang, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No